CLINICAL TRIAL: NCT03235869
Title: A Single Arm Pilot Study of Radiation Therapy Plus Durvalumab for Tumor-Stage Cutaneous T-Cell Lymphoma
Brief Title: Radiation Therapy Plus Durvalumab for Tumor-Stage Cutaneous T-Cell Lymphoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The company pulled durvalumab from heme malignancies
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.079; HUM00131550 (Other: University of Michigan)
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Radiation Therapy + Durvalumab (Experimental): Radiation to 1-3 cutaneous tumors: 20 Gy (4 Gy x 5 fractions) Durvalumab 1500mg IV over 1 hour administered within 2-7 days of initiation of radiation, then every 28 days.
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg IV over 1 hour administered within 2-7 days of initiation of radiation, then every 28 days.
Radiation: Radiation Therapy — Radiation to 1-3 cutaneous tumors: 20 Gy (4 Gy x 5 fractions)

SUMMARY:
This is a single arm, single stage pilot study of radiation therapy plus durvalumab for tumor-stage cutaneous T-cell lymphoma (CTCL).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily provide written IRB-approved consent
* Age ≥ 18 years
* Histologically proven CTCL
* Stage IIB-IV CTCL with ≥2 cutaneous tumors assessable for response
* At least one cutaneous tumor amenable to radiation therapy. Must have at least 1 tumor assessable for response that will not undergo radiation.
* Adequate organ function
* Prior treatment is allowed if at least 4 weeks have elapsed since last chemotherapy and/or radiation and the subject has recovered from all treatment related toxicity

Exclusion Criteria:

* Prior allogeneic stem cell transplant.
* Prior treatment with a PD-1/PD-L1 inhibitor
* Active or prior documented autoimmune or inflammatory disorders within the past 3 years prior to the start of treatment.
* Current or prior use of immunosuppressive medication within 14 days prior to first dose of durvalumab.
* Known human immunodeficiency virus (HIV), hepatitis C virus (HCV) or active hepatitis B virus (HBV) infection.
* History of hypersensitivity to durvalumab or any excipient
* Receipt of live attenuated vaccination within 30 days prior the first dose of durvalumab.
* Female subjects who are pregnant, breast-feeding or female patients of reproductive potential who are not employing an effective method of birth control
* Male subjects who are not employing an effective method of birth control
* Uncontrolled current medical illness, including, but not limited to ongoing or active infections, symptomatic congestive heart failure, unstable angina pectoris,unstable cardiac arrhythmia and/or psychiatric illness or other condition that in the opinion of the investigator would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients that respond to treatment | 1 year post treatment
  Overall Response Rate (ORR) is defined as the percentage of patients that obtain a Complete Response (CR) or Partial Response (PR) to treatment. A global composite scoring system will be used to determine response. Skin, nodes, viscera and blood will be assessed.
The percentage of patients that completely respond to treatment | 1 year post treatment
  Complete Response Rate (CRR) is defined as the percentage of patients that obtain Complete Response (CR) to treatment. A global composite scoring system will be used to determine response. Skin, nodes, viscera and blood will be assessed.

SECONDARY OUTCOMES:
Time to response | 1 year post treatment
  The time to response is measured from the start of the treatment until criteria are met for CR or PR. A global composite scoring system will be used to determine response. Skin, nodes, viscera and blood will be assessed.
Duration of overall response | 1 year post treatment
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrence or PD (Progressive disease) is objectively documented. A global composite scoring system will be used to determine response and progression. Skin, nodes, viscera and blood will be assessed.
Progression free survival time | 1 year post treatment
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death. A global composite scoring system will be used to determine progression. Skin, nodes, viscera and blood will be assessed.
Time to next treatment | 1 year post treatment
  Time to next treatment is defined as the duration of time from start of study treatment to next treatment or death of any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: "Ryan Wilcox, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States